CLINICAL TRIAL: NCT05141955
Title: A Randomized Controlled Trial for Postoperative Analgesia in Patients Undergoing Laparoscopic Sleeve Gastrectomy: Ultrasound Guided Erector Spinae Plane Block Versus Quadratus Lumborum Block
Brief Title: Ultrasound Guided Erector Spinae Plane Block Versus Quadratus Lumborum Block for Postoperative Analgesia in Patients Undergoing Laparoscopic Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dr.Ibrahim Mamdouh Esmat, Assistant Professor of Anesthesia and Intensive Care Department, Faculty of Medicine, Ain- shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU MS 705/ 2021
Record Dates: First submitted 2021-11-30; First posted 2021-12-02 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Population Groups; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Erector Spinae Plane Block (ESPB) (Active Comparator)
  Interventions: Other: Group Erector Spinae Plane Block (ESPB)
- Group Quadratus Lumborum Block (QLB) (Active Comparator)
  Interventions: Other: Group Quadratus Lumborum Block (QLB)
- Group (C) (Control group) (Other)
  Interventions: Other: Group (C) (Control group)

INTERVENTIONS:
Other: Group Erector Spinae Plane Block (ESPB) — Patients will receive general anesthesia initially then bilateral ESPB with a total volume of (0.3-0.4 ml/kg LBW) of bupivacaine 0.25% will be performed (not exceeding toxic dose) 150 mg "
  Arms: Group Erector Spinae Plane Block (ESPB)
Other: Group Quadratus Lumborum Block (QLB) — Patients will receive general anesthesia initially then bilateral QLB with a total volume of (0.3-0.4 ml/kg LBW) of bupivacaine 0.25% will be performed "not exceeding toxic dose150 mg "
  Arms: Group Quadratus Lumborum Block (QLB)
Other: Group (C) (Control group) — Where patients will be operated under general anesthesia.
  Arms: Group (C) (Control group)

SUMMARY:
Postoperative pain control is a signiﬁcant challenge in medical practice. Inadequate pain control could decrease patient's satisfaction, delay postoperative ambulation, increase the incidence of pulmonary and cardiac complications and cause the development of chronic postoperative pain. Laparoscopic surgical techniques could decrease postoperative pain and opioid consumption.

The addition of regional techniques to general anesthesia showed better pain management and less consumption of opioids compared to the traditional techniques.

The aim of this study is to compare the effectiveness of ultrasound guided erector spinae plane block versus quadratus lumborum block regarding postoperative analgesia in patients undergoing laparoscopic sleeve gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with free medical history or controlled hypertension and/ or diabetes scheduled for elective laparoscopic sleeve gastrectomy.
* BMI > 35 kg/ m2

Exclusion Criteria:

* Patients unfit for surgery or refuse to sign the consent of regional block.
* Patients with known coagulation defects.
* Patients with known hypersensitivity to bupivacaine.
* Patients with infection at the site of injection.
* Conversion of laparoscopic surgery to laparotomy

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Time to first requested rescue analgesia(Minutes) | 24 hours postoperatively
  Time to first requested rescue analgesia(Minutes)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain-Shams University Hospitals, Cairo, Egypt